CLINICAL TRIAL: NCT03582033
Title: A Phase 1 Study of SEA-BCMA in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Safety Study of SEA-BCMA in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNBCMA-001
Record Dates: First submitted 2018-06-12; First posted 2018-07-10 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: RRMM; Antibodies, monoclonal; Antigens, BCMA; Immunotherapy; Hematologic diseases; Myeloma; Seattle Genetics
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases; Neoplasms, Plasma Cell | interventions — Dexamethasone; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Parts A and B: SEA-BCMA Monotherapy (Experimental): SEA-BCMA
  Interventions: Drug: SEA-BCMA
- Part C: SEA-BCMA + Dexamethasone Combination Therapy (Experimental): SEA-BCMA + dexamethasone
  Interventions: Drug: SEA-BCMA; Drug: dexamethasone
- Part D: SEA-BCMA + Pomalidomide + Dexamethasone Combination Therapy (Experimental): SEA-BCMA + dexamethasone + pomalidomide
  Interventions: Drug: SEA-BCMA; Drug: dexamethasone; Drug: pomalidomide

INTERVENTIONS:
Drug: SEA-BCMA — Given into the vein (IV; intravenously)
Drug: dexamethasone — Given by mouth (orally) or by IV
  Arms: Part C: SEA-BCMA + Dexamethasone Combination Therapy; Part D: SEA-BCMA + Pomalidomide + Dexamethasone Combination Therapy
Drug: pomalidomide — Given orally
  Arms: Part D: SEA-BCMA + Pomalidomide + Dexamethasone Combination Therapy

SUMMARY:
This trial will study SEA-BCMA to find out whether it is an effective treatment for multiple myeloma (MM) and what side effects (unwanted effects) may occur.

The study will have several parts. In Parts A and B, participants get SEA-BCMA by itself. This part of the study will find out how much SEA-BCMA should be given for treatment and how often. It will also find out how safe the treatment is and how well it works.

In Part C of the study, participants will get SEA-BCMA and dexamethasone. In Part D, participants will get SEA-BCMA, dexamethasone, and pomalidomide. Dexamethasone and pomalidomide are both drugs that can be used to treat multiple myeloma. These parts of the study will find out whether these drugs are safe when used together.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of MM
* Must have MM that is relapsed or refractory
* Has received a proteasome inhibitor, an immunomodulatory drug, and an anti-CD38 antibody
* Measurable disease, as defined by at least one of the following: (1) serum M protein 0.5 g/dL or higher, (2) urine M protein 200 mg/24 hour or higher, and (3) serum immunoglobulin free light chain (FLC) 10 mg/dL or higher and abnormal serum immunoglobulin kappa lambda FLC ratio.
* Eastern Cooperative Oncology Group (ECOG) status score of 0 or 1
* Life expectancy of greater than 3 months in the opinion of the investigator
* Adequate hematologic, renal, and hepatic function

Exclusion Criteria:

* Parts A and D: Prior treatment with a BCMA-directed therapy
* History of another malignancy within 3 years
* Active cerebral or meningeal disease related to the underlying malignancy
* Uncontrolled Grade 3 or higher infection
* Prior antitumor therapy that is not completed at least 4 weeks prior to first dose of study drug, or at least 2 weeks if progressing. Prior CAR-T-cell therapy must be completed 8 weeks before first dose of study drug.
* Combination therapy only:

  1. Known intolerance to corticosteroids
  2. Uncontrolled psychoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hayman, MD, Study Director — Seagen Inc.
Locations (13):
- United States (13):
  - Stanford University School of Medicine, Palo Alto, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Holden Comprehensive Cancer Center / University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Washington University in St Louis, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - James P. Wilmot Cancer Center / University of Rochester Medical Center, Rochester, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 106 participants signed the informed consent form. 15 participants were screen failures, 8 were not assigned to receive study treatment and 83 participants received at least 1 dose of study treatment.
Pre-assignment Details: This study had following parts: Part A (SEA-[B-cell maturation antigen] BCMA) monotherapy, Part B (SEA-BCMA monotherapy intensive dosing), Part C (SEA-BCMA and dexamethasone combination) and Part D (SEA-BCMA, pomalidomide and dexamethasone combination).
Groups:
- Part A: SEA-BCMA 100mg: Participants received SEA-BCMA 100 milligrams (mg) as a monotherapy once every 2 weeks (q2wk) intravenous (IV) on Day 1 and 15 of each 28- day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part A: SEA-BCMA 200mg: Participants received SEA-BCMA 200 mg as a monotherapy q2wk IV on Day 1 and 15 of each 28- day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part A: SEA-BCMA 400mg: Participants received SEA-BCMA 400 mg as a monotherapy q2wk IV on Day 1 and 15 of each 28- day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part A: SEA-BCMA 800mg: Participants received SEA-BCMA 800 mg as a monotherapy q2wk IV on Day 1 and 15 of each 28- day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part A: SEA-BCMA 1600mg: Participants received SEA-BCMA 1600 mg as a monotherapy q2wk IV on Day 1 and 15 of each 28- day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part B: SEA-BCMA 1600mg: Participants received SEA-BCMA 1600 mg as an IV infusion once every 1 week (q1wk) as induction dose for the first two cycles, followed by q2wk as maintenance dose in subsequent cycles, of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part C: SEA-BCMA 1600mg and Dexamethasone: Participants received SEA-BCMA 1600 mg IV q2wk on Day 1 and 15 of each 28-day cycle, and dexamethasone 40 mg orally or as an IV infusion on Day 1, 8, 15, and 22 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part C: SEA-BCMA 800mg and Dexamethasone: Participants received SEA-BCMA 800 mg IV q1wk on Day 1 and 15 of each 28-day cycle, and dexamethasone 40 mg orally or as an IV infusion on Day 1, 8, 15, and 22 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part C: SEA-BCMA 1600 mg and Dexamethasone: Participants received SEA-BCMA 1600 mg IV q1wk on Day 1,8,15 and 22 of each 28-day cycle, and dexamethasone 40 mg orally or as an IV infusion on Day 1, 8, 15, and 22 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone: Participants received SEA-BCMA 1600 mg IV q2wk on Day 1 and 15 of each 28-day cycle, dexamethasone 40 mg orally or as an IV infusion on Day 1, 8, 15, and 22 and pomalidomide 4 mg orally, daily from Day 1 to 21 of each of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
Period: Part A
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg | Part B: SEA-BCMA 1600mg | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Started | 2 | 2 | 2 | 7 | 22 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 2 | 7 | 22 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 2 | 4 | 11 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg | Part B: SEA-BCMA 1600mg | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Started | 0 | 0 | 0 | 0 | 0 | 20 (Participants who were enrolled in Part-B of the study.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Period: Part C
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg | Part B: SEA-BCMA 1600mg | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Started | 0 | 0 | 0 | 0 | 0 | 0 | 12 (Participants who were enrolled in Part-C of the study.) | 6 (Participants who were enrolled in Part-C of the study.) | 5 (Participants who were enrolled in Part-C of the study.) | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 6 | 5 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 2 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Period: Part D
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg | Part B: SEA-BCMA 1600mg | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 (Participants who were enrolled in Part-D of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Groups:
- Part A: SEA-BCMA 100mg: Participants received SEA-BCMA 100 mg as a monotherapy q2wk IV on Day 1 and 15 of each 28- day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Part B: SEA-BCMA 1600mg: Participants received SEA-BCMA 1600 mg as an IV infusion q1wk as induction dose for the first two cycles, followed by q2wk as maintenance dose in subsequent cycles, of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurs first.
- Total: Total of all reporting groups
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg | Part B: SEA-BCMA 1600mg | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone | Total
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22 | 20 | 12 | 6 | 5 | 5 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (2.1) | 70.0 (7.1) | 72.5 (9.2) | 64.3 (10.6) | 73.3 (7.9) | 73.2 (8.9) | 66.9 (8.5) | 74.3 (6.5) | 72.6 (3.9) | 71.2 (6.6) | 71.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 2 | 10 | 7 | 7 | 2 | 2 | 2 | 36
  Male | 0 | 2 | 0 | 5 | 12 | 13 | 5 | 4 | 3 | 3 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 1 | 1 | 9
  Not Hispanic or Latino | 2 | 2 | 2 | 6 | 18 | 19 | 10 | 5 | 4 | 4 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3 | 1 | 2 | 3 | 0 | 1 | 0 | 13
  White | 0 | 1 | 2 | 4 | 19 | 17 | 9 | 6 | 3 | 5 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), Treatment Related TEAEs and Greater Than or Equal to (>=) Grade 3 TEAEs: Part A
Description: An adverse event (AE) was any untoward medical occurrence in a participant/ clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs were defined as newly occurring (not present at baseline)/worsening after first dose of investigational product (IP). TESAEs were any untoward medical occurrence at any dose that: suspected to cause death; life-threatening; required hospitalization; persistent/significant disability/incapacity & may cause congenital anomaly/birth defect. Treatment related TEAEs were related to study treatment and relatedness was judged by investigator. TEAEs were graded according to National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (v) 4.03 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening).
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment up to 44 months (maximum follow up of 45 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Participants
  TEAEs | 2 | 2 | 2 | 6 | 20
  TESAEs | 1 | 1 | 2 | 3 | 8
  Treatment Related TEAEs | 0 | 0 | 1 | 4 | 13
  TEAEs (>= Grade 3) | 1 | 1 | 2 | 4 | 13

2. Primary Outcome: Number of Participants With TEAEs, TESAEs, Treatment Related TEAEs and >=Grade 3 TEAEs: Part B
Description: An AE was any untoward medical occurrence in a participant/ clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs were defined as newly occurring (not present at baseline)/worsening after first dose of IP. TESAEs were any untoward medical occurrence at any dose that: suspected to cause death; life-threatening; required hospitalization; persistent/significant disability/incapacity & may cause congenital anomaly/birth defect. Treatment related TEAEs were related to study treatment and relatedness was judged by investigator. TEAEs were graded according to NCI CTCAE v 4.03 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening).
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment up to 33 months (maximum follow up of 34 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 20
Participants
  TEAEs | 19
  TESAEs | 5
  Treatment Related TEAEs | 7
  TEAEs (>= Grade 3) | 6

3. Primary Outcome: Number of Participants With TEAEs, TESAEs, Treatment Related TEAEs and >=Grade 3 TEAEs: Part C
Description: as for outcome 2
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment up to 36 months (maximum follow up of 37 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 6 | 5
Participants
  TEAEs | 11 | 6 | 5
  TESAEs | 5 | 3 | 2
  Treatment Related TEAEs | 4 | 0 | 3
  TEAEs (>= Grade 3) | 8 | 5 | 3

4. Primary Outcome: Number of Participants With TEAEs, TESAEs, Treatment Related TEAEs and >=Grade 3 TEAEs: Part D
Description: as for outcome 2
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment up to 19 months (maximum follow up of 20 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 5
Participants
  TEAEs | 5
  TESAEs | 3
  Treatment Related TEAEs | 3
  TEAEs (>= Grade 3) | 3

5. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Serum Chemistry: Part A
Description: The following serum chemistry laboratory parameters were assessed: Alanine aminotransferase high, albumin low, alkaline phosphatase high, amylase high, aspartate aminotransferase high, calcium corrected for albumin high, calcium corrected for albumin low, creatinine high, glucose high, glucose low, lipase high, phosphate low, potassium high, potassium low, sodium high, sodium low, total bilirubin high and urate high. Chemistry laboratory parameters abnormalities were graded according to NCI CTCAE v 4.03 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Participants with any serum chemistry parameter meeting CTCAE grade 1 to 4 were reported.
Time Frame: as for outcome 1
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Participants
  Grade 1 | 0 | 1 | 0 | 1 | 4
  Grade 2 | 0 | 0 | 0 | 3 | 7
  Grade 3 | 0 | 1 | 2 | 2 | 11
  Grade 4 | 2 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Serum Chemistry: Part B
Description: as for outcome 5
Time Frame: as for outcome 2
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 20
Participants
  Grade 1 | 5
  Grade 2 | 8
  Grade 3 | 6
  Grade 4 | 1

7. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Serum Chemistry: Part C
Description: as for outcome 5
Time Frame: as for outcome 3
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 6 | 5
Participants
  Grade 1 | 0 | 1 | 1
  Grade 2 | 5 | 1 | 2
  Grade 3 | 5 | 3 | 2
  Grade 4 | 2 | 1 | 0

8. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Serum Chemistry: Part D
Description: as for outcome 5
Time Frame: as for outcome 4
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 5
Participants
  Grade 1 | 1
  Grade 2 | 1
  Grade 3 | 3
  Grade 4 | 0

9. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Hematology: Part A
Description: The following hematology laboratory parameters were assessed: hemoglobin high, hemoglobin low, leukocytes high, leukocytes low, lymphocytes high, lymphocytes low, neutrophils low and platelets low. Laboratory abnormality events were graded according to NCI CTCAE v 4.03 (grade 1=mild, grade 2=moderate, grade 3= severe and grade 4= life-threatening). Participants with any hematology parameter meeting CTCAE grade 1 to 4 were reported.
Time Frame: as for outcome 1
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Participants
  Grade 1 | 0 | 1 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 1 | 12
  Grade 3 | 1 | 1 | 1 | 4 | 9
  Grade 4 | 1 | 0 | 0 | 2 | 1

10. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Hematology: Part B
Description: as for outcome 9
Time Frame: as for outcome 2
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 20
Participants
  Grade 1 | 6
  Grade 2 | 6
  Grade 3 | 7
  Grade 4 | 1

11. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Hematology: Part C
Description: as for outcome 9
Time Frame: as for outcome 3
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 6 | 5
Participants
  Grade 1 | 1 | 1 | 1
  Grade 2 | 3 | 3 | 0
  Grade 3 | 4 | 2 | 3
  Grade 4 | 4 | 0 | 1

12. Primary Outcome: Number of Participants With Maximum Laboratory Toxicity Grade, by NCI-CTCAE v4.03- Hematology: Part D
Description: as for outcome 9
Time Frame: as for outcome 4
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 5
Participants
  Grade 1 | 0
  Grade 2 | 2
  Grade 3 | 1
  Grade 4 | 2

13. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs): Part A
Description: The DLT-evaluation period was the first cycle of treatment. DLTs were graded according to the NCI-CTCAE, v 4.03, and were defined as any of the following events during the DLT-evaluation period: a ) A delay of SEA-BCMA treatment by more than 7 days due to toxicity, b) Any AE >=Grade 3, unless deemed by the safety monitoring committee (SMC) to be clearly unrelated to SEA-BCMA except for the AEs as pre specified in protocol to be considered a DLT and c) Any treatment related death.
Time Frame: Cycle 1 (28 days)
Population: The DLT-evaluable (DE) analysis set included treated participants who either experienced a DLT, or were followed up for the full DLT evaluation period and received at least 75% of the intended total Cycle 1 SEA-BCMA dose, and did not receive prohibited treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 7
Participants | 0 | 0 | 0 | 1 | 0

14. Primary Outcome: Number of Participants With DLTs: Part B
Description: The DLT-evaluation period was the first cycle of treatment. DLTs were graded according to the NCI-CTCAE, v 4.03, and were defined as any of the following events during the DLT-evaluation period: a ) A delay of SEA-BCMA treatment by more than 7 days due to toxicity, b) Any AE >=Grade 3, unless deemed by the SMC to be clearly unrelated to SEA-BCMA except for the AEs as pre specified in protocol to be considered a DLT and c) Any treatment related death.
Time Frame: Cycle 1 (28 days)
Population: The DE analysis set included treated participants who either experienced a DLT, or were followed up for the full DLT evaluation period and received at least 75% of the intended total Cycle 1 SEA-BCMA dose, and did not receive prohibited treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 6
Participants | 0

15. Primary Outcome: Number of Participants With DLTs: Part C
Description: as for outcome 14
Time Frame: Cycle 1 (28 days)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 4 | 5 | 4
Participants | 0 | 0 | 0

16. Primary Outcome: Number of Participants With DLTs: Part D
Description: as for outcome 14
Time Frame: Cycle 1 (28 days)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 4
Participants | 0

17. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Day 14 (AUC0-14) of SEA-BCMA: Part A
Description: Area under the observed concentration-time curve from the time of dosing to Day 14 calculated by log-linear trapezoidal approximation.
Time Frame: Cycle 1 and 2: Pre dose, 1 and 2 hour intradose, end of drug administration, 2, 6 , 24, 72, 168 and 336 hours post end of infusion on Day 1
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter (ug/mL)
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Day*micrograms per milliliter (ug/mL)
  Cycle 1 | 181.3 (20.0) | 302.6 (14.6) | 977.2 (37.0) | 1443.2 (23.9) | 3267.7 (26.8)
  Cycle 2: number analyzed (Participants) | 2 | 2 | 1 | 6 | 12
  Cycle 2 | 244.8 (15.4) | 436.0 (10.6) | 2216.4 (NA) — Geometric Coefficient of variation (CV) could not be calculated as only 1 participant was available for analysis. | 2387.9 (41.4) | 5972.1 (61.0)

18. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Day 7 (AUC0-7) of SEA-BCMA: Part A
Description: Area under the observed concentration-time curve from the time of dosing to Day 7 calculated by log-linear trapezoidal approximation.
Time Frame: Cycle 1: Pre dose, 1 and 2 hour intradose, end of drug administration, 2, 6 , 24, 72, and 168 hours post end of infusion on Day 1
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ug/mL
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Day*ug/mL | 112.6 (17.6) | 197.6 (11.1) | 626.5 (26.3) | 932.0 (22.1) | 2064.5 (23.4)

19. Secondary Outcome: AUC0-7 of SEA-BCMA: Part B
Description: as for outcome 18
Time Frame: as for outcome 18
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ug/mL
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 7
Day*ug/mL | 2001.3 (26.4)

20. Secondary Outcome: AUC0-7 of SEA-BCMA: Part C
Description: as for outcome 18
Time Frame: as for outcome 18
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ug/mL
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 3 | 2
Day*ug/mL | 2011.8 (32.9) | 840.3 (21.2) | 1629.3 (20.9)

21. Secondary Outcome: AUC0-7 of SEA-BCMA: Part D
Description: as for outcome 18
Time Frame: as for outcome 18
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ug/mL
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 1
Day*ug/mL | 1926.2 (NA) — Geometric CV could not be calculated as only 1 participant was available for analysis.

22. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of SEA-BCMA: Part A
Time Frame: Cycle 1 and 2: Pre dose, 1 and 2 hour intradose, end of drug administration, 2, 6 , 24, 72, 168 and 336 hours post end of infusion on Day 1 and 15
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (ug/mL)
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 21
Micrograms per milliliter (ug/mL)
  Cycle 1 | 28.5 (32.3) | 47.2 (3.9) | 134.8 (11.6) | 236.4 (14.4) | 494.6 (20.3)
  Cycle 2: number analyzed (Participants) | 2 | 1 | 1 | 6 | 16
  Cycle 2 | 44.9 (3.6) | 62.4 (NA) — Geometric CV could not be calculated as only 1 participant was available for analysis. | 213.1 (NA) — Geometric CV could not be calculated as only 1 participant was available for analysis. | 307.4 (34.1) | 746.6 (29.7)

23. Secondary Outcome: Cmax of SEA-BCMA: Part B
Time Frame: Cycle 1: Pre dose, 1 and 2 hour intradose, end of drug administration, 2, 6 , 24, 72, 168 and 336 hours post end of infusion on Day 1 and 15
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 19
ug/mL | 493.3 (27.7)

24. Secondary Outcome: Cmax of SEA-BCMA: Part C
Time Frame: as for outcome 23
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 5 | 4
ug/mL | 471.5 (72.3) | 204.2 (27.3) | 486.4 (17.9)

25. Secondary Outcome: Cmax of SEA-BCMA: Part D
Time Frame: Cycle 1:Pre dose, 1 and 2 hour intradose, end of drug administration, 2, 6 , 24, 72, 168 and 336 hours post end of infusion on Day 1 and 15
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 4
ug/mL | 415.1 (31.8)

26. Secondary Outcome: Number of Participants With SEA-BCMA Antitherapeutic Antibodies (ATA): Part A
Description: A positive baseline ATA result was considered positive post-baseline if the post-baseline ATA titer result was at least four times higher than the baseline result.
Time Frame: Anytime during study (maximum up to 45 months)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 1 | 7 | 21
Participants | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With SEA-BCMA, ATA: Part B
Description: as for outcome 26
Time Frame: Anytime during study (maximum up to 34 months)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 17
Participants | 0

28. Secondary Outcome: Number of Participants With SEA-BCMA, ATA: Part C
Description: as for outcome 26
Time Frame: Anytime during study (maximum up to 37 months)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 3 | 5
Participants | 0 | 0 | 0

29. Secondary Outcome: Number of Participants With SEA-BCMA, ATA: Part D
Description: as for outcome 26
Time Frame: Anytime during study (maximum up to 20 months)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 2
Participants | 0

30. Secondary Outcome: Objective Response Rate (ORR) as Per the International Myeloma Working Group (IMWG) Uniform Response Criteria: Part A
Description: ORR: Percentage of participants with an objective response (OR) per investigator. Participant was determined to have an OR if, based on 2016 IMWG uniform response criteria, & achieved stringent complete response (sCR), Complete response (CR), very good partial response(VGPR) & partial response(PR): free light chain(FLC) ratio & absence of clonal cells in bone marrow by immunohistochemistry(IC)/ immunofluorescence(IF). CR: negative immunofixation of serum & urine, disappearance of any soft tissue plasmacytomas(STP), 5% plasma cells in bone marrow. VGPR: serum & urine M-protein (UMP) detectable by immunofixation but not on electrophoresis/ >= 90% reduction in serum M-protein (SMP) level+UMP level <100 mg/24 hr, PR: >=50% reduction of SMP & reduction in 24-hr urinary M-protein by >=90%/to <200 mg/24 hr. If SMP & UMP are unmeasurable, a ≥50% decrease in the difference between involved & uninvolved FLC levels were required in place of the M-protein criteria.
Time Frame: From the first dose of study treatment until the first documented sCR or CR or PR or VGPR or new anti-cancer therapies or death, whichever occurred first (maximum up to 45 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 41.0] | 14 [2.9 to 34.9]

31. Secondary Outcome: ORR as Per the IMWG Uniform Response Criteria: Part B
Description: The ORR was defined as the percentage of participants with an OR per investigator. A participant was determined to have an OR if, based on the 2016 IMWG uniform response criteria, and achieved a sCR, CR, VGPR, or a PR. sCR: FLC ratio & absence of clonal cells in bone marrow by IC/IF. CR: negative immunofixation of serum & urine, disappearance of any STP, 5% plasma cells in bone marrow. VGPR: serum and UMP detectable by immunofixation but not on electrophoresis or >= 90% reduction in SMP level+UMP level <100 mg/24 hour, PR: >=50% reduction of SMP & reduction in 24-hour urinary M-protein by >=90%/to <200 mg/24 hour. If SMP & UMP are unmeasurable, a ≥50% decrease in the difference between involved & uninvolved FLC levels were required in place of the M-protein criteria. In addition to above criteria, if present at baseline, >=50% reduction in the size of STP were also required.
Time Frame: From the first dose of study treatment until the first documented sCR or CR or PR or VGPR or new anti-cancer therapies or death, whichever occurred first (maximum up to 34 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 20
Percentage of participants | 20 [5.7 to 43.7]

32. Secondary Outcome: ORR as Per the IMWG Uniform Response Criteria: Part C
Description: as for outcome 31
Time Frame: From the first dose of study treatment until the first documented sCR or CR or PR or VGPR or new anti-cancer therapies or death, whichever occurred first (maximum up to 37 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 6 | 5
Percentage of participants | 17 [2.1 to 48.4] | 33 [4.3 to 77.7] | 20 [0.5 to 71.6]

33. Secondary Outcome: ORR as Per the IMWG Uniform Response Criteria: Part D
Description: The ORR was defined as the percentage of participants with an OR per investigator. A participant was determined to have an OR if, based on the 2016 IMWG uniform response criteria, and achieved a sCR, CR, VGPR, or a PR. sCR: FLC ratio & absence of clonal cells in bone marrow by IC/IF. CR: negative immunofixation of serum & urine, disappearance of any STP, 5% plasma cells in bone marrow. VGPR: serum and UMP detectable by immunofixation but not on electrophoresis/ >= 90% reduction in SMP level+UMP level <100 mg/24 hour, PR: >=50% reduction of SMP & reduction in 24-hour urinary M-protein by >=90%/to <200 mg/24 hour. If SMP & UMP are unmeasurable, a ≥50% decrease in the difference between involved & uninvolved FLC levels were required in place of the M-protein criteria. In addition to above criteria, if present at baseline, >=50% reduction in the size of STP were also required.
Time Frame: From the first dose of study treatment until the first documented sCR or CR or PR or VGPR or new anti-cancer therapies or death, whichever occurred first (maximum up to 20 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 5
Percentage of participants | 80 [28.4 to 99.5]

34. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) as Per the IMWG Uniform Response Criteria: Part A
Description: BOR consisted of MRD-negative CR,sCR,CR,VGPR,PR,MR,SD & PD per 2016 IMWG. MRD: evaluated using adaptive next generation sequencing(NGS) for MRD assay & carried out on relevant specimen to understand activity of SEA-BCMA. sCR: CR & normal FLC ratio & absence of clonal cells in bone marrow by IC/ IF. CR: Negative immunofixation of serum & urine disappearance of any STP, & <5% plasma cells in bone marrow. VGPR: SMP & UMP detectable by IF but not on electrophoresis/ >= 90% reduction(R) in SMP level+UMP level <100 mg/24 hr, PR: >=50% R of SMP & R in 24-hr UMP by >=90%/by <200 mg/24 hr. If SMP & UMP are unmeasurable, >=50% decrease in difference between involved & uninvolved FLC levels were required in place of M-protein criteria. SD: Not meeting criteria for CR, VGPR, PR, MR, or progression. MR: 25-49% R of SMP & R in 24-hr UMP by 50-89%, which still exceeds 200mg/24 hr. DP: objective evidence of tumor progression(based on serum/urine/BM assessments) &/clinical progression/investigator.
Time Frame: as for outcome 30
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Percentage of participants
  Minimal Residual Disease (MRD)-negative complete response (CR) | 0 | 0 | 0 | 0 | 0
  Stringent complete response (sCR) | 0 | 0 | 0 | 0 | 0
  Complete response (CR) | 0 | 0 | 0 | 0 | 0
  Very good partial response (VGPR) | 0 | 0 | 0 | 0 | 5
  Partial response (PR) | 0 | 0 | 0 | 0 | 9
  Minimal response (MR) | 0 | 0 | 0 | 0 | 5
  Stable disease (SD) | 50 | 100 | 0 | 86 | 45
  Progressive disease (DP) | 50 | 0 | 100 | 14 | 36

35. Secondary Outcome: Percentage of Participants With BOR as Per the IMWG Uniform Response Criteria: Part B
Description: BOR consisted of MRD-negative CR, sCR, CR, VGPR, PR, MR, SD & PD per 2016 IMWG. MRD: evaluated using adaptive NGS for MRD assay & carried out on relevant specimen to understand activity of SEA-BCMA. sCR: CR & normal FLC ratio & absence of clonal cells in bone marrow by IC/ IF. CR: Negative immunofixation of serum & urine disappearance of any STP, & <5% plasma cells in bone marrow. VGPR: SMP & UMP detectable by IF but not on electrophoresis/ >= 90% reduction(R) in SMP level+UMP level <100 mg/24 hr, PR: >=50% R of SMP & R in 24-hr UMP by >=90%/by <200 mg/24 hr. If SMP & UMP are unmeasurable, >=50% decrease in difference between involved & uninvolved FLC levels were required in place of M-protein criteria. SD: Not meeting criteria for CR, VGPR, PR, MR, or progression. MR: 25-49% R of SMP & R in 24-hr UMP by 50-89%, which still exceeds 200mg/24 hr. DP: objective evidence of tumor progression(based on serum/urine/BM assessments) &/clinical progression/investigator.
Time Frame: as for outcome 31
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number; unit: Percentage of participants
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 20
Percentage of participants
  MRD-negative CR | 0
  sCR | 5
  CR | 0
  VGPR | 0
  PR | 15
  MR | 5
  SD | 55
  DP | 15

36. Secondary Outcome: Percentage of Participants With BOR as Per the IMWG Uniform Response Criteria: Part C
Description: BOR consisted of MRD-negative CR, sCR, CR, VGPR, PR, MR, SD & PD per 2016 IMWG. MRD: evaluated using NGS for MRD assay & carried out on relevant specimen to understand activity of SEA-BCMA. sCR: CR & normal FLC ratio & absence of clonal cells in bone marrow by IC/ IF. CR: Negative immunofixation of serum & urine disappearance of any STP, & <5% plasma cells in bone marrow. VGPR: SMP & UMP detectable by IF but not on electrophoresis/ >= 90% reduction(R) in SMP level+UMP level <100 mg/24 hr, PR: >=50% R of SMP & R in 24-hr UMP by >=90%/by <200 mg/24 hr. If SMP & UMP are unmeasurable, >=50% decrease in difference between involved & uninvolved FLC levels were required in place of M-protein criteria. SD: Not meeting criteria for CR, VGPR, PR, MR, or progression. MR: 25-49% R of SMP & R in 24-hr UMP by 50-89%, which still exceeds 200mg/24 hr. DP: objective evidence of tumor progression(based on serum/urine/BM assessments) &/clinical progression/investigator.
Time Frame: as for outcome 32
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number; unit: Percentage of participants
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 6 | 5
Percentage of participants
  MRD-negative CR | 0 | 0 | 0
  sCR | 8 | 0 | 0
  CR | 0 | 0 | 0
  VGPR | 0 | 17 | 0
  PR | 8 | 17 | 20
  MR | 0 | 17 | 0
  SD | 67 | 33 | 60
  DP | 17 | 17 | 20

37. Secondary Outcome: Percentage of Participants With BOR as Per the IMWG Uniform Response Criteria: Part D
Description: BOR consisted of MRD-negative CR,sCR,CR,VGPR,PR,MR,SD & PD per 2016 IMWG. MRD: evaluated using adaptive NGS for MRD assay & carried out on relevant specimen to understand activity of SEA-BCMA. sCR: CR & normal FLC ratio & absence of clonal cells in bone marrow by IC/ IF. CR: Negative immunofixation of serum & urine disappearance of any STP, & <5% plasma cells in bone marrow. VGPR: SMP & UMP detectable by IF but not on electrophoresis/ >= 90% reduction(R) in SMP level+UMP level <100 mg/24 hr, PR: >=50% R of SMP & R in 24-hr UMP by >=90%/by <200 mg/24 hr. If SMP & UMP are unmeasurable, >=50% decrease in difference between involved & uninvolved FLC levels were required in place of M-protein criteria. SD: Not meeting criteria for CR, VGPR, PR, MR, or progression. MR: 25-49% R of SMP & R in 24-hr UMP by 50-89%, which still exceeds 200mg/24 hr. DP: objective evidence of tumor progression(based on serum/urine/BM assessments) &/clinical progression/investigator.
Time Frame: as for outcome 33
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Number; unit: Percentage of participants
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 5
Percentage of participants
  MRD-negative CR | 0
  sCR | 40
  CR | 0
  VGPR | 20
  PR | 20
  MR | 0
  SD | 20
  DP | 0

38. Secondary Outcome: Duration of Objective Response (DOR) as Per the IMWG Uniform Response Criteria: Part A
Description: DOR: Time from first documentation of OR(sCR,CR,VGPR/PR) to first documentation of PD/death due to any cause, whichever came first. PD: Objective evidence of tumor progression(TP) (based on serum, urine/BM assessments) &/clinical progression/ investigator. sCR: CR, normal FLC ratio & absence of clonal cells in bone marrow by IC/IF. CR: Negative immunofixation of serum&urine, disappearance of any STP, &<5% plasma cells in bone marrow. VGPR: Serum & UMP detectable by immunofixation but not on electrophoresis/ >= 90% reduction(R) in SMP level+UMP level <100 mg/24 hour, PR: >=50%R of SMP & R in 24-hour UMP by >=90% or to <200 mg/24 hour. DOR: censored on date of last disease assessment documenting absence of PD for participants who do not have PD & were still on study at the time of an analysis/removed from study prior to documentation of TP. Participants started new antitumor treatment prior to documentation of PD were censored at last disease assessment prior to start of new treatment.
Time Frame: From the first dose of study treatment until the first documented OR (sCR or CR or PR or VGPR) on or before the first documented PD or death or censoring date, whichever occurred first (maximum up to 45 months)
Population: as for outcome 19
Measure: Median (Full Range); unit: Months
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Months |  |  |  |  | 10.0 [5.5 to 15.2]

39. Secondary Outcome: DOR as Per the IMWG Uniform Response Criteria: Part B
Description: as for outcome 38
Time Frame: From the first dose of study treatment until the first documented OR (sCR or CR or PR or VGPR) on or before the first documented PD or death or censoring date, whichever occurred first (maximum up to 34 months)
Population: as for outcome 19
Measure: Median (Full Range); unit: Months
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 4
Months | 8.4 [1.8 to 31.5]

40. Secondary Outcome: DOR as Per the IMWG Uniform Response Criteria: Part C
Description: as for outcome 38
Time Frame: From the first dose of study treatment until the first documented OR (sCR or CR or PR or VGPR) on or before the first documented PD or death or censoring date, whichever occurred first (maximum up to 37 months)
Population: as for outcome 19
Measure: Median (Full Range); unit: Months
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 2 | 2 | 1
Months | NA [4.6 to 35.7] — Median could not be calculated due to insufficient number of participants with events. | NA [1.9 to 22.6] — Median could not be calculated due to insufficient number of participants with events. | 6.5 [6.5 to 6.5]

41. Secondary Outcome: DOR as Per the IMWG Uniform Response Criteria: Part D
Description: as for outcome 38
Time Frame: From the first dose of study treatment until the first documented OR (sCR or CR or PR or VGPR) on or before the first documented PD or death or censoring date, whichever occurred first (maximum up to 20 months)
Population: as for outcome 19
Measure: Median (Full Range); unit: Months
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 4
Months | 8.3 [2.6 to 18.9]

42. Secondary Outcome: Progression Free Survival (PFS): Part A
Description: PFS: Time from the start of any study treatment to first documentation of DP or to death due to any cause, whichever comes first. DP included objective evidence of tumor progression (based on serum, urine or BM assessments) and/or clinical progression per investigator. PFS was censored on the date of the last disease assessment documenting absence of PD for participants who do not have disease progression and are still on study at the time of an analysis, or discontinuation of study prior to documentation of tumor progression. Participants who have started a new antitumor treatment prior to documentation of PD were censored at the last disease assessment prior to start of new treatment. Participants lacking an evaluation of tumor response after their first dose had their event time censored as 1 day.
Time Frame: From the date of first dose until the first documentation of PD or death or censoring date, whichever occurred first (maximum up to 45 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Months | 1.7 [0.7 to 2.8] | 5.9 [0.7 to 11.0] | 0.7 [0.7 to 0.7] | 4.4 [0.6 to 15.5] | 2.1 [0.5 to 42.9]

43. Secondary Outcome: PFS: Part B
Description: as for outcome 42
Time Frame: From the date of first dose until the first documentation of PD or death or censoring date, whichever occurred first (maximum up to 34 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 20
Months | 1.7 [0.5 to 33.1]

44. Secondary Outcome: PFS: Part C
Description: as for outcome 42
Time Frame: From the date of first dose until the first documentation of PD or death or censoring date, whichever occurred first (maximum up to 37 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 6 | 5
Months | 1.6 [0.7 to 36.4] | 3.2 [0.7 to 24.1] | 3.5 [0.7 to 7.2]

45. Secondary Outcome: PFS: Part D
Description: as for outcome 42
Time Frame: From the date of first dose until the first documentation of PD or death or censoring date, whichever occurred first (maximum up to 20 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 5
Months | 10.1 [1.8 to 19.6]

46. Secondary Outcome: Overall Survival (OS): Part A
Description: OS was defined as the time from the start of any study treatment to the date of death due to any cause. OS was calculated as date of death minus date of first dose of any study treatment plus 1. OS for participants who were alive at their date of last contact, including those lost to follow-up, were censored at the date of last contact. If the last recorded date where a participant was known to be alive is the date of first dose of any study treatment, survival time was censored on the date of first dose of any study treatment (i.e., OS duration of 1 day).
Time Frame: From date of start of study treatment until date of death or censoring date (maximum up to 45 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 22
Months | 9.2 [3.0 to 9.2] | 37.5 [11.1 to 37.5] | 8.1 [0.9 to 15.3] | 19.2 [1.3 to 45.3] | 19.7 [0.9 to 44.3]

47. Secondary Outcome: OS: Part B
Description: as for outcome 46
Time Frame: From date of start of study treatment until date of death or censoring date (maximum up to 34 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B: SEA-BCMA 1600mg
Number analyzed (Participants) | 20
Months | NA [0.8 to 33.7] — Median could not be calculated due to insufficient number of participants with events.

48. Secondary Outcome: OS: Part C
Description: as for outcome 46
Time Frame: From date of start of study treatment until date of death or censoring date (maximum up to 37 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone
Number analyzed (Participants) | 12 | 6 | 5
Months | 18.0 [1.9 to 36.4] | NA [3.7 to 26.0] — Median could not be calculated due to insufficient number of participants with events. | 12.2 [1.2 to 22.2]

49. Secondary Outcome: OS: Part D
Description: as for outcome 46
Time Frame: From date of start of study treatment until date of death or censoring date (maximum up to 20 months)
Population: All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Measure: Median (Full Range); unit: Months
Arm/Group | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
Number analyzed (Participants) | 5
Months | NA [3.3 to 19.6] — Median could not be calculated due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment for Part A: up to 44 months (maximum follow up of 45 months); Part B: up to 33 months (maximum follow up of 34 months); Part C: up to 36 months (maximum follow up of 37 months) and Part D: up to 19 months (maximum follow up of 20 months)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. All treated participants analysis set included all treated participants who received any amount of SEA-BCMA.
Arm/Group | Part A: SEA-BCMA 100mg | Part A: SEA-BCMA 200mg | Part A: SEA-BCMA 400mg | Part A: SEA-BCMA 800mg | Part A: SEA-BCMA 1600mg | Part B: SEA-BCMA 1600mg | Part C: SEA-BCMA 1600mg and Dexamethasone | Part C: SEA-BCMA 800mg and Dexamethasone | Part C: SEA-BCMA 1600 mg and Dexamethasone | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/2 | 2/2 | 4/7 | 11/22 | 2/20 | 6/12 | 1/6 | 2/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 2/2 | 3/7 | 8/22 | 5/20 | 5/12 | 3/6 | 2/5 | 3/5
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 6/7 | 18/22 | 17/20 | 10/12 | 5/6 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: SEA-BCMA 100mg (N=2) | Part A: SEA-BCMA 200mg (N=2) | Part A: SEA-BCMA 400mg (N=2) | Part A: SEA-BCMA 800mg (N=7) | Part A: SEA-BCMA 1600mg (N=22) | Part B: SEA-BCMA 1600mg (N=20) | Part C: SEA-BCMA 1600mg and Dexamethasone (N=12) | Part C: SEA-BCMA 800mg and Dexamethasone (N=6) | Part C: SEA-BCMA 1600 mg and Dexamethasone (N=5) | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: SEA-BCMA 100mg (N=2) | Part A: SEA-BCMA 200mg (N=2) | Part A: SEA-BCMA 400mg (N=2) | Part A: SEA-BCMA 800mg (N=7) | Part A: SEA-BCMA 1600mg (N=22) | Part B: SEA-BCMA 1600mg (N=20) | Part C: SEA-BCMA 1600mg and Dexamethasone (N=12) | Part C: SEA-BCMA 800mg and Dexamethasone (N=6) | Part C: SEA-BCMA 1600 mg and Dexamethasone (N=5) | Part D: SEA-BCMA 1600 mg, Pomalidomide and Dexamethasone (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid haematoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (2) | 1 (1) | 3 (3) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 8 (9) | 7 (8) | 6 (6) | 1 (1) | 2 (2) | 2 (3)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 4 (6) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (3)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 3 (5) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunoglobulins decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (4) | 2 (4) | 2 (2) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 2 (2) | 3 (4) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (4) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain fog (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jugular vein occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyarteritis nodosa (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03582033/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT03582033/SAP_001.pdf